CLINICAL TRIAL: NCT02646072
Title: The Effect of Preoperative Topical Ketorolac 0.45% on Aqueous Cytokine Levels and Macular Thickness in Diabetic and Non Diabetic Patients Undergoing Cataract Surgery
Brief Title: Effect of Preoperative Topical Ketorolac on Aqueous Cytokine Levels and Macular Thickness in Cataract Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Lai Yin Peng, MD, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20148-494
Record Dates: First submitted 2015-12-12; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Cystoid Macular Edema, Postoperative; Diabetes Mellitus
Keywords: diabetes mellitus; aqueous humor; inflammatory cytokines; cystoid macular edema, postoperative; nonsteroidal anti-inflammatory drugs
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diabetes mellitus patients (Active Comparator): Ketorolac tromethamine ophthalmic solution 0.45% four times a day for 3 days prior to cataract surgery
  Interventions: Drug: Ketorolac tromethamine ophthalmic solution 0.45%
- Diabetes mellitus control patients (No Intervention): Topical refresh plus four times a day for 3 days prior to cataract surgery
- Non diabetic patients (Active Comparator): Ketorolac tromethamine ophthalmic solution 0.45% four times a day for 3 days prior to cataract surgery
  Interventions: Drug: Ketorolac tromethamine ophthalmic solution 0.45%
- Non diabetic control patients (No Intervention): Topical refresh plus four times a day for 3 days prior to cataract surgery

INTERVENTIONS:
Drug: Ketorolac tromethamine ophthalmic solution 0.45% — Indicated for the treatment of pain and inflammation following cataract surgery.
  Other Names: Acuvail
  Arms: Diabetes mellitus patients; Non diabetic patients

SUMMARY:
The purpose of this study is to determine whether there is a relationship between inflammatory cytokines in the aqueous of the eye and thickness of the macula after treatment of topical ketorolac for patients undergoing cataract surgery.

DETAILED DESCRIPTION:
To compare aqueous levels of inflammatory cytokines in diabetic and non diabetic patients treated with preoperative topical ketorolac tromethamine 0.45%.

To compare the macular thickness changes in diabetic and non diabetic patients treated with preoperative ketorolac tromethamine 0.45% and its correlation with the aqueous inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

Diabetic patient group

1. Type 2 diabetes mellitus with no diabetic retinopathy
2. If with co-morbid, controlled hypertension with no hypertensive crisis in recent six months
3. Listed for phacoemulsification cataract surgery

Non diabetic patient group

1. No history of diabetes
2. If with co-morbid, controlled hypertension with no hypertensive crisis in recent six months
3. Listed for phacoemulsification cataract surgery

Exclusion Criteria:

1. Smoker
2. Presence of immune disease, local or systemic inflammation
3. Presence of retinal diseases, glaucoma
4. Previous surgical procedure on the eye
5. Intra-operative complications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Level of aqueous inflammatory cytokines post treatment as assessed using Bio-plex Pro Assays | 9 months
  Aqueous samples were analyzed at the same after complete samples collection.

SECONDARY OUTCOMES:
Changes from baseline in central subfield retinal thickness as assessed by optical coherence tomography | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Yin Peng Lai, MOphthal, Principal Investigator — University of Malaya; Mohammadreza Peyman, Mophthal, Study Chair — University of Malaya; Tajunisah Iqbal, FRCS Ophth, Study Director — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheung CM, Vania M, Ang M, Chee SP, Li J. Comparison of aqueous humor cytokine and chemokine levels in diabetic patients with and without retinopathy. Mol Vis. 2012;18:830-7. Epub 2012 Apr 4. PMID 22511846
- [Background] Dong N, Xu B, Wang B, Chu L. Study of 27 aqueous humor cytokines in patients with type 2 diabetes with or without retinopathy. Mol Vis. 2013 Aug 4;19:1734-46. Print 2013. PMID 23922491
- [Background] Chu L, Wang B, Xu B, Dong N. Aqueous cytokines as predictors of macular edema in non-diabetic patients following uncomplicated phacoemulsification cataract surgery. Mol Vis. 2013 Nov 24;19:2418-25. eCollection 2013. PMID 24319335
- [Background] Yilmaz T, Cordero-Coma M, Gallagher MJ. Ketorolac therapy for the prevention of acute pseudophakic cystoid macular edema: a systematic review. Eye (Lond). 2012 Feb;26(2):252-8. doi: 10.1038/eye.2011.296. Epub 2011 Nov 18. PMID 22094296
- [Background] Schoenberger SD, Kim SJ, Sheng J, Calcutt MW. Reduction of vitreous prostaglandin E2 levels after topical administration of ketorolac 0.45%. JAMA Ophthalmol. 2014 Feb;132(2):150-4. doi: 10.1001/jamaophthalmol.2013.5692. PMID 24264034
- [Background] Schoenberger SD, Kim SJ, Shah R, Sheng J, Cherney E. Reduction of interleukin 8 and platelet-derived growth factor levels by topical ketorolac, 0.45%, in patients with diabetic retinopathy. JAMA Ophthalmol. 2014 Jan;132(1):32-7. doi: 10.1001/jamaophthalmol.2013.6203. PMID 24336915
- [Background] Henderson BA, Kim JY, Ament CS, Ferrufino-Ponce ZK, Grabowska A, Cremers SL. Clinical pseudophakic cystoid macular edema. Risk factors for development and duration after treatment. J Cataract Refract Surg. 2007 Sep;33(9):1550-8. doi: 10.1016/j.jcrs.2007.05.013. PMID 17720069
- [Background] Almeida DR, Johnson D, Hollands H, Smallman D, Baxter S, Eng KT, Kratky V, ten Hove MW, Sharma S, El-Defrawy S. Effect of prophylactic nonsteroidal antiinflammatory drugs on cystoid macular edema assessed using optical coherence tomography quantification of total macular volume after cataract surgery. J Cataract Refract Surg. 2008 Jan;34(1):64-9. doi: 10.1016/j.jcrs.2007.08.034. PMID 18165083
- [Background] Wittpenn JR, Silverstein S, Heier J, Kenyon KR, Hunkeler JD, Earl M; Acular LS for Cystoid Macular Edema (ACME) Study Group. A randomized, masked comparison of topical ketorolac 0.4% plus steroid vs steroid alone in low-risk cataract surgery patients. Am J Ophthalmol. 2008 Oct;146(4):554-560. doi: 10.1016/j.ajo.2008.04.036. Epub 2008 Jul 2. PMID 18599019
- [Background] Bucci FA Jr, Waterbury LD. A randomized comparison of to-aqueous penetration of ketorolac 0.45%, bromfenac 0.09% and nepafenac 0.1% in cataract patients undergoing phacoemulsification. Curr Med Res Opin. 2011 Dec;27(12):2235-9. doi: 10.1185/03007995.2011.626018. Epub 2011 Oct 12. PMID 21992076
- [Background] Heier JS, Awh CC, Busbee BG, Waterbury LD, Daniel P, Stoller GL, Cleary TS. Vitreous nonsteroidal antiinflammatory drug concentrations and prostaglandin E2 levels in vitrectomy patients treated with ketorolac 0.4%, bromfenac 0.09%, and nepafenac 0.1%. Retina. 2009 Oct;29(9):1310-3. doi: 10.1097/IAE.0b013e3181b094e6. PMID 19934822
- [Background] Ozturk BT, Bozkurt B, Kerimoglu H, Okka M, Kamis U, Gunduz K. Effect of serum cytokines and VEGF levels on diabetic retinopathy and macular thickness. Mol Vis. 2009 Sep 19;15:1906-14. PMID 19784389
- [Background] Hanifi-Moghaddam P, Kappler S, Seissler J, Muller-Scholze S, Martin S, Roep BO, Strassburger K, Kolb H, Schloot NC. Altered chemokine levels in individuals at risk of Type 1 diabetes mellitus. Diabet Med. 2006 Feb;23(2):156-63. doi: 10.1111/j.1464-5491.2005.01743.x. PMID 16433713
- [Background] Oh IK, Kim SW, Oh J, Lee TS, Huh K. Inflammatory and angiogenic factors in the aqueous humor and the relationship to diabetic retinopathy. Curr Eye Res. 2010 Dec;35(12):1116-27. doi: 10.3109/02713683.2010.510257. PMID 21121809
- [Background] Bressler NM, Edwards AR, Antoszyk AN, Beck RW, Browning DJ, Ciardella AP, Danis RP, Elman MJ, Friedman SM, Glassman AR, Gross JG, Li HK, Murtha TJ, Stone TW, Sun JK; Diabetic Retinopathy Clinical Research Network. Retinal thickness on Stratus optical coherence tomography in people with diabetes and minimal or no diabetic retinopathy. Am J Ophthalmol. 2008 May;145(5):894-901. doi: 10.1016/j.ajo.2007.12.025. Epub 2008 Feb 21. PMID 18294608
- [Background] Gharbiya M, Cruciani F, Cuozzo G, Parisi F, Russo P, Abdolrahimzadeh S. Macular thickness changes evaluated with spectral domain optical coherence tomography after uncomplicated phacoemulsification. Eye (Lond). 2013 May;27(5):605-11. doi: 10.1038/eye.2013.28. Epub 2013 Mar 1. PMID 23449512